CLINICAL TRIAL: NCT00270244
Title: Group Interpersonal Psychotherapy for Depressed Adolescents (IPT-AG) in School-based Clinics
Brief Title: Group Interpersonal Psychotherapy for Depressed Adolescents in School-based Clinics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01 MH73640, #5037; R01MH073640 (NIH); DSIR 84-CTS
Record Dates: First submitted 2005-12-21; First posted 2005-12-26 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Depression
Keywords: Major Depression; Dysthymic Disorder; Adjustment Disorder With Depressed Mood; Depressive Disorder Not Otherwise Specified; Adolescent; Psychotherapy
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Dysthymic Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Participants will receive treatment as usual
  Interventions: Behavioral: Treatment as usual (TAU)
- 2 (Experimental): Participants will receive group interpersonal psychotherapy for depressed adolescents
  Interventions: Behavioral: Group interpersonal psychotherapy for depressed adolescents (IPT-AG)

INTERVENTIONS:
Behavioral: Group interpersonal psychotherapy for depressed adolescents (IPT-AG) — Participants assigned to IPT-AG will attend two to three, 40-minute individual pre-group sessions, followed by 12, 90-minute group therapy sessions and two additional individual sessions-one midway through the group sessions and another upon completion of group therapy. Sessions will focus on problems in interpersonal relationships.
  Arms: 2
Behavioral: Treatment as usual (TAU) — TAU will consist of counseling sessions as regularly conducted by the school clinic social worker and/or referral to another agency.
  Arms: 1

SUMMARY:
This study will assess the effectiveness of group interpersonal psychotherapy (IPT-AG) versus treatment as usual (TAU) in improving the treatment of depressed adolescents in school-based health clinics.

DETAILED DESCRIPTION:
Depression is a serious medical condition. It occurs in people of all ages, but only in the past two decades has depression in children and adolescents been taken seriously. Children and adolescents with depression may exhibit such behaviors as pretending to be sick, refusing to go to school or getting in trouble at school, clinging to a parent or worrying that the parent may die, sulking, or acting in a negative or grouchy manner. A previous study demonstrated that, when administered by clinicians in school-based clinics, individual interpersonal psychotherapy is effective in reducing depressive symptoms and improving global and social functioning. This study will assess the effectiveness of group interpersonal psychotherapy (IPT-AG) versus treatment as usual (TAU) in improving depressive symptoms of adolescents in school-based health clinics.

Participants in this 16-week single-blind study will be randomly assigned to receive either IPT-AG or TAU in a school-based clinic. Participants assigned to receive IPT-AG will attend two to three, 40-minute individual pre-group sessions, followed by 12, 90-minute group therapy sessions and two additional individual sessions-one midway through the group sessions and another upon completion of group therapy. TAU will consist of counseling sessions as regularly conducted by the school clinic social worker and/or referral to another agency. Study visits will occur at baseline and Weeks 4, 8, 12, and 16, or upon early termination. At the end of 16 weeks, participants assigned to receive IPT-AG will continue in a maintenance program in which they will receive IPT-AG once a month for an additional 6 months. All participants will also be assessed 6 and 12 months post-treatment to measure depressive symptoms, global and social functioning, satisfaction with care, and utilization of other services.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for major depression, dysthymic disorder, depressive disorder not otherwise specified, or adjustment disorder with depressed mood
* Score of 24 or greater on the CES-D
* Score between 10 and 28 on the HRSD
* Score of 65 or less on the C-GAS
* English-speaking
* Parental or legal guardian consent to participate

Exclusion Criteria:

* Actively suicidal
* Score greater than 28 on the HRSD
* Mentally retarded
* Any life threatening medical illness
* Meets diagnostic criteria for current substance abuse, schizophrenia, or bipolar disorder
* Any evidence of psychosis, conduct disorder, or active eating disorder
* Currently in active treatment for depression
* Taking antidepressant medication at the time of baseline assessment
* Recent death of someone close

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2005-12; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms as measured by the Hamilton Rating Scale for Depression (HRSD) and the Center for Epidemiological Studies-Depression Scale (CES-D) | Measured at Month 18
Overall impairment, as measured by the Global Assessment Scale for Children (C-GAS) | Measured at Month 18
Social functioning, as measured by the Social Adjustment Scale-Self-report (SAS-SR) | Measured at Month 18

SECONDARY OUTCOMES:
Short Acculturation Scale for Hispanics, CES-D, HRSD, C-GAS, Clinical Global Improvement, Inventory of Parent and Peer Attachment, Family Adaptation and Cohesions Evaluation Scales III, and the Penn Helping Alliance Questionnaire-Revised | Measured at Month 18

CONTACTS AND LOCATIONS:
Overall Officials: Laura H. Mufson, PhD, Principal Investigator — New York State Psychiatric Institute-Columbia University College of Physicians and Surgeons